CLINICAL TRIAL: NCT05607784
Title: An Interactive Education Program to Reduce High Risk Behavior in Adolescents Ph I
Brief Title: Education Program to Reduce Risky Behavior in Adolescents Ph I
Acronym: iTRAC
Status: Completed | Type: Observational
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: Rhode Island Hospital (Other); University of Oregon (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0342; 1R42HD110333-01 (NIH)
Record Dates: First submitted 2022-10-13; First posted 2022-11-07 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Risky Sexual Behavior; Emotional Regulation; Adolescent Behavior
MeSH Terms: conditions — Emotional Regulation; Adolescent Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescent Advisory Board Male: This board consisted of 9 male adolescents recruited from the schools.
  Interventions: Behavioral: Formative Research- Content Translation
- Adolescent Advisory Board Female: This board consisted of 9 female adolescents recruited from the schools.
  Interventions: Behavioral: Formative Research- Content Translation
- Health Education Professionals Panel (HEPP): This panel consisted of 6 health teachers and other school health professionals such as nurses and counselors. They were recruited at each participating school.
  Interventions: Behavioral: Formative Research- Content Feedback and Acceptability

INTERVENTIONS:
Behavioral: Formative Research- Content Translation — This formative research includes brainstorming translation of content and reviewing wireframe prototypes generated from this process. It also includes attending to cultural, developmental, and gender considerations.
  The design development cycles will begin with advisory focus group feedback about how the existing activities convey the content (i.e., what and how they are learning). They will advise on activity design for the remaining content (sexual health and content connecting this with ER) to ensure these are engaging, appropriate, and informative. They will also provide perspectives about design, structure, navigability, and approach
  Groups: Adolescent Advisory Board Female; Adolescent Advisory Board Male
Behavioral: Formative Research- Content Feedback and Acceptability — This formative research includes providing feedback on the proposed content and ensure contextual acceptability in schools.
  The design development cycles will begin with advisory focus group feedback about how the existing activities convey the content (i.e., what and how they are learning). They will advise on activity design for the remaining content (sexual health and content connecting this with ER) to ensure these are engaging, appropriate, and informative. They will also provide perspectives about design, structure, navigability, and approach
  Groups: Health Education Professionals Panel (HEPP)

SUMMARY:
This phase will complete the TRAC adaptation to a web app. The pilot study (R21 HD089979) effectively translated the ER content of TRAC and the same procedures will be used to translate the remaining content.

DETAILED DESCRIPTION:
Adolescence is a critical developmental period during which behavioral patterns are formed that have powerful influences on current and future health. This is particularly true for sexual behavior, which is affected by the bio-logical changes of puberty as well as normative developmental tasks around sexual exploration. Engaging in sexual behavior in early adolescence (before age 15) is associated with more partners, less condom use, and more frequent sex as teens get older, and these factors increase risk for negative health outcomes (e.g., sexually transmitted infections and unplanned pregnancy) throughout their lives. Many sexual health interventions teach prevention skills, such as assertiveness or condom use; the premise of the current application is that these skills are often unused by adolescents because of deficits in emotion regulation (ER), which is un-addressed in most sexual health education. The research team has developed and tested a novel, engaging, efficacious, and developmentally tailored group intervention (Project TRAC) to teach ER skills to early adolescents within the context of sexual health. A study of Project TRAC showed that participants taught ER skills were less likely to start having sex over the 2.5 year follow up. While efficacious, the small group format of the program presents barriers to sustainability and dissemination; significant advantages of web-based delivery exist. To explore whether the ER concepts of TRAC could be taught in a web-based format, the investigators completed a pilot study to translate TRAC's ER content to a web-based intervention (iTRAC), using Designing for Dissemination principles that enhance the likelihood of successful dissemination upon completion. iTRAC demonstrated feasibility and acceptability, and a randomized trial showed that iTRAC participants reported significantly better emotional competence compared to waitlist control participants. The proposed Fast Track project will complete the technology adaptation of the program to include its sexual health content and content linking ER to sexual health. This adaptation (iTRAC for Sexual Risk Prevention; iTRAC-SRP), using well-established theoretical frameworks, will be approached with advisory boards of school professionals and early adolescents, leading to prototypes of the completed intervention in Phase 1.

ELIGIBILITY:
Inclusion Criteria for Adolescent Advisory Boards:

* Attending 7th grade
* Between 12 and 14 years old
* Parent/guardian speaks English or Spanish
* Attending participating school

Exclusion Criteria for Adolescent Advisory Boards:

* Unable to read at a 4th grade level
* Have a sibling who has participated in the study
* Have a developmental disorder

Inclusion Criteria for Health Education Professionals:

* Work at participating schools
* Directly involved in the health of middle school students
* Adult (at least 18)

Exclusion Criteria for Health Education Professionals:

* Teachers not directly involved in the health of middle school students

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The adolescent advisory board members and the health education professionals will be recruited from participating schools.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Formative Research | Baseline, After wireframe production (approximately 2 months after baseline)
  Advisory Focus Groups: Research summaries will also be generated to communicate with participating communities. Using these recommended D4D processes, the research will be better positioned for dissemination (and commercialization)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Houck, PhD, Principal Investigator — Rhode Island Hospital
Locations (3):
- United States (3):
  - Klein Buendel, Golden, Colorado
  - University of Oregon, Eugene, Oregon
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
The investigators will prepare an archival-quality data package for upload to the National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH). Specifically, the investigators will provide documentation on the full data-audit trail from the exact prompts seen by participants, to the syntax used to score and aggregate items, to the finalized data ready for use by qualified investigators. The archival-quality data package will also include a codebook in line with the Data Documentation Initiative (DDI) and contains information about variables, metadata, and file structure. The metadata will include description of the trial, including design, implementation, and description of the interventions. The intent is to provide everything that future investigators require to understand the trial, analyze the data, correctly interpret the findings, and be able to publish new analyses that meet current publication standards for clinical trials and/or meta-analyses.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After analyses are completed for the aims of the study
Access Criteria: The data package will be available for future investigators. For datasets that include potentially sensitive information, investigators not part of the original study will submit requests to be reviewed by the PIs. Qualified investigators who agree to terms of use and confidentiality agreements will be provided with deidentified data.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT05607784/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT05607784/ICF_001.pdf